Statistical Analysis Plan


# SAFETY AND EFFICACY OF CD5024 0.3% CREAM IN SUBJECTS WITH ATOPIC DERMATITIS

## STATISTICAL ANALYSIS PLAN RD.03.SPR.109696

13 JULY 2017

This document is electronically approved and signed by: Statistic Manager

Name PPD Reason for Signing PPD

Date 21-Jul-2017


| A | | +1 | • | 01 |
|---|---|----|---|----|
| | u | u | ш | |

PPD

Responsible of the statistical analysis

Reviewer:

PPD PPD

Statistical Analysis Plan 

# **DOCUMENT HISTORY**

| Version No. | Description of Edits | Justification | Date |
|---|---|---|---|
| Amendment 1 | The analysis of the primary endpoint changes from the percent change in EASI score from baseline to week 6 to the Change in EASI score from baseline to week 6 adjusted on baseline. Change from baseline will be analyzed on ITT-LOCF, ITT-MI and PP. As a secondary endpoint Percentage change in EASI score from baseline to any scheduled visits will be analyzed via a Cochran Mantel Haenszel test stratified by analysis center, using RIDIT transformation and Row mean score statistics. Percent change from baseline will be analyzed on ITT-LOCF and PP | distribution and for the intended analysis (ANOVA) increases the residual error and thus makes the statistical test less powerful and not appropriate. | |

Statistical Analysis Plan 

# TABLE OF CONTENTS

| 1 | STUDY OBJECTIVES6 |
|---|---|
| 2 | STUDY DESIGN6 |
| 3 | EFFICACY AND SAFETY VARIABLES8 |
| 3.1 | Efficacy variables8 |
| 3.1.1 | Primary efficacy endpoints8 |
| 3.1.2 | Secondary efficacy endpoints8 |
| 4 | SAFETY AND OTHER VARIABLES8 |
| CCI | 8 |
| 5 | POPULATIONS ANALYZED9 |
| 5.1 | Intent-to-treat (ITT) Efficacy analysis set9 |
| 5.2 | Per-protocol (PP) Efficacy analysis set9 |
| 5.3 | Safety population9 |
| 5.4 | PK set9 |
| 6 | SAMPLE SIZE CONSIDERATION10 |
| 7 | STATISTICAL METHODS AND DATA CONSIDERATIONS10 |
| 7.1 | Study subjects |
| 7.1.1 | Disposition of subjects10 |
| 7.1.2 | Protocol deviations10 |
| 7.2 | Efficacy analysis |
| 7.2.1 | Data sets analyzed11 |
| 7.2.2 | Demographic and baseline characteristics11 |
| 7.2.3 | Medical history, previous and concomitant therapies and previous and concomitant procedures11 |
| 7.2.4 | Compliance11 |
| 7.2.5 | Statistical analysis for efficacy12 |
| 7.2.6 | Statistical and analytical issues13 |
| 7.3 | Safety analysis14 |
| 7.3.1 | Extent of exposure14 |

Statistical Analysis Plan 

| CCI | | 15 |
|---|---|---|
| 7.3.3 | Laboratory parameters | 15 |
| 7.3.4 | Vital signs, physical findings and other observations related to safety | 15 |
| CCI | | 16 |
| | | 16 |
| | | 16 |
| 7.5 | Analysis visit definition | 16 |
| 8 | CHANGES FROM THE PROTOCOL ANALYSIS PLAN | 17 |
| 9 | TABLES, FIGURES, AND GRAPHS | 17 |
| 9.1 | Study subject | 17 |
| 9.2 | Efficacy analysis | 23 |
| 9.2.1 | Primary efficacy endpoint | 23 |
| 9.2.2 | Secondary efficacy endpoints | 32 |
| 9.2.3 | Subgroup analyses | 44 |
| 9.3 | Safety analysis | 46 |
| 9.3.1 | Extent of exposure | 46 |
| CCI | | 47 |
| 9.3.3 | Laboratory parameters | 50 |
| 9.3.4 | Vital Sign and physical examination and other information related to safety | 55 |
| CCI | | 57 |

Statistical Analysis Plan


#### 1 STUDY OBJECTIVES

The primary objective of this study is to evaluate the local and systemic safety of CD5024 0.3% cream applied once daily over a 6-week treatment period in adults with chronic lesions of moderate atopic dermatitis (AD), compared to its vehicle.

The secondary objective is to evaluate the efficacy of CD5024 0.3 % cream versus its vehicle on chronic lesions of moderate AD.

CCI

#### 2 STUDY DESIGN

This is an exploratory, multi-center (approximately 5 sites in Canada), randomized, vehicle-controlled, investigator-blind, parallel group study, involving approximately 85 subjects screened to get approximately 60 randomized subjects with chronic lesions of AD meeting specific inclusion/non-inclusion criteria. The investigator and/or other evaluator(s) will not come into contact with the study materials. Subjects and the study staff do not have access to the correspondence between the kit number and the assigned treatment group.

Subjects who consent to be enrolled and fulfill study criteria will be allocated to one of the study treatment according to the randomization list, in a 1:1 ratio (for example Group A: N=30 subjects treated with CD5024 0.3% cream, and Group B: N=30 subjects treated with the vehicle).

Statistical Analysis Plan


## Efficacy and safety assessments

| | Screening<br>period | | | | | | Treat | ment | Period | | | | | | Early<br>Termina | Unsche<br>duled | Follow<br>-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week-5 to<br>Week-1 | W | eek 1 | We | eek 2 | W | eek 3 | We | eek 4 | k4 We | | We | ek 6 | Week<br>7 | tion | | Week<br>9 |
| | D-30 to D-3 | D01 | D02 to<br>D07 | D0 8 | D09 to<br>D14 | D15 | D16 to<br>D21 | D22 | D23 to<br>D28 | D29 | D30 to<br>D35 | D36 | D37 to<br>D42 | D43 | | | D54±2 |
| Efficacy assessment | | | | | | | | | | | | | | | | | |
| EASI Score | | Х | | Х | | Х | | Х | | Х | | X | | X (b) | X | X | |
| Investigator Global Assessment (IGA) | Х | Х | | Х | | Х | | Х | | Х | | Х | | X (b) | Х | | |
| TSS | | Х | | Х | | Х | | Х | | Х | | X | | X (b) | Х | | |
| Modified-Objective SCORAD | | Х | | Х | | Х | | Х | | Х | | X | | X (b) | Х | | |
| Hand IGA when applicable | | Х | | Х | | Х | | Х | | Х | | Х | | X (b) | Х | | |
| tBSA (Total Body Surface Area) | Х | | | | | | | | | | | | | | | | |
| BSA (i.e. affected by AD) | Х | Х | | Х | | Х | | Х | | Х | | X | | X (b) | Х | X | |
| Patient-reported Outcome - Pruritus Numerical<br>Rating Scale & DIARY | х | Х | Х | Х | Х | X | X | X | Х | X | X | X | Х | X (b) | Х | | |
| Patient-reported Outcome - Pruritus Verbal<br>Rating Scale & DIARY | | Х | | | | | | | | | | | | X (b) | х | | |
| Safety assessment | | | | | | | | | | | | | | | | | |
| Blood samplings (coagulation, hematology, biochemistry) | х | | | | | | | X | | | | | | Х | х | | |
| Blood samplings (IgE & TARC) | Х | | | | | | | | | | | | | Х | Х | | |
| Physical examination | X | Х | | | | Х | | | | Х | | | | Х | Х | | X |
| Vital signs | X | Х | | | | Х | | | | Х | | | | Х | Х | | Х |
| ECG | X | Х | | | | | | | | | | | | Х | Х | | |
| CCI | | | | | | | | | | | | | | | | | |
| Other assessment | | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | |

CCI

(b) All assessments are to be done before any procedures are performed.

Statistical Analysis Plan


#### 3 EFFICACY AND SAFETY VARIABLES

### 3.1 Efficacy variables

#### 3.1.1 Primary efficacy endpoints

The Primary efficacy endpoint is the change from Baseline to Week 6 of the EASI score.

## 3.1.2 Secondary efficacy endpoints

The change from Baseline of the EASI score at any other evaluation visit and the percent change from Baseline in EASI score at each evaluation visit.

Investigator Global Assessment in terms of distribution and in terms of success rate (success is defined as a subject with an IGA score of 0 [clear] or 1 [Almost clear]) at each evaluation visit.

Percent change from Baseline of the Total Sum Score (TSS) of the target plaque.

Change from Baseline of each individual score (Erythema, Induration/Papulation, Oozing/Crusting, Excoriation, Lichenification).

Percent Change from baseline of the Modified Objective SCORAD.

Pruritus (numerical rating scale [NRS], verbal rating scale [VRS]) and their changes from Baseline at each evaluation visit.

#### 4 SAFETY AND OTHER VARIABLES

Physical examination, Vital signs (pulse rate and blood pressure)

Laboratory parameters

Adverse events



Statistical Analysis Plan


#### 5 POPULATIONS ANALYZED

## 5.1 Intent-to-treat (ITT) Efficacy analysis set

The ITT set is defined as any subjects who are randomized. Data from subjects included in the ITT population will be analyzed according to the treatment as randomized.

## 5.2 Per-protocol (PP) Efficacy analysis set

The PP set is defined as the ITT population, after exclusion of subjects deemed non-evaluable for efficacy due to major deviations from the protocol. Major deviations are divided into 4 categories:

- Entrance criteria deviations,
- Non-compliance,
- Concomitant therapies taken during the study and/or Concomitant illnesses, interfering with efficacy,
- Administrative errors such as unblinding or study drug dispensing errors.

Major deviations will be identified and categorized before database lock and unblinding, during a blind data review meeting.

## 5.3 Safety population

The Safety set is defined as comprising the ITT Population subjects who applied/were administered the study drug(s) at least once. In practice, only the subjects who return their study drug(s) unopened will be excluded from the Safety Population. All safety data will be summarized based on the Safety Population.

#### **5.4 PK** set

The PK set is defined as comprising all subjects from the safety set who have signed the ICF for PK samples and who provide at least one post-baseline evaluable drug concentration value. All PK data will be based on observed cases.


#### **6 SAMPLE SIZE CONSIDERATION**

In a previous Galderma R&D trial (SPR.18158) where a Vehicle was used in atopic dermatitis in subjects with involved BSA between 5% and 20%, the Vehicle percent change from Baseline at Week 4 of a modified EASI (No Head and Neck) was -40% and the standard deviation (SD) was 45%.

In studies evaluating Dupilumab versus placebo, the observed placebo EASI score percent changes from Baseline at Week 4 ranged from -17% to -25% with a SD around 40% (Beck 2014), and was - 18% at Week 16 with a standard deviation of 40% (Thaci 2016). In this last trial it was observed that these values were reached from week 4 onwards. Based on these historical data, the SD was set at 40%.

The magnitude of effect of Dupilumab reached 45% over placebo. However, systemic immunosuppressant drug for atopic dermatitis are generally more effective than topical treatments (Thaci 2016). Taking that into account, for CD5024 cream 0.3% applied once daily, an effect of 30% over its vehicle would be considered as clinically relevant. Consequently, the effect size (delta/sigma) has been set at 0.75 (30%/40%).

Using a randomization ratio of 1:1 for CD5024 cream 0.3% QD and vehicle, a sample size of 30 randomized subjects in each treatment group can ensure an 80% power to detect a difference of 30 % between CD5024 and its vehicle on EASI score mean percent change from Baseline.

## 7 STATISTICAL METHODS AND DATA CONSIDERATIONS

For statistical analyses purpose, baseline is defined as the last measurement prior to the first application of the study drug. This is true for all variables except NRS, for which baseline is the mean of the values collected from Day -3 to Day -1.

## 7.1 Study subjects

#### 7.1.1 Disposition of subjects

Reasons for early discontinuation, and normal completions, will be summarized using frequency distribution (n, %).

#### 7.1.2 Protocol deviations

Major protocol deviations will be summarized overall using frequency distribution (n, %).


## 7.2 Efficacy analysis

#### 7.2.1 Data sets analyzed

Number of subjects included in each efficacy analyses (ITT, PP) and number of subjects included in the safety analysis will be presented by treatment.

## 7.2.2 Demographic and baseline characteristics

The subject demographics and baseline characteristics will be summarized by descriptive statistics.

- Frequency distribution (n, %), for qualitative criteria,
- Usual statistics (n, mean, standard deviation, median, min, max), for quantitative criteria,
- Both frequency distribution and usual statistics for ordinal criteria.

# 7.2.3 Medical history, previous and concomitant therapies and previous and concomitant procedures

Frequency distribution of subjects with at least one previous or/and concomitant disease at inclusion will be given.

Previous and Concomitant therapies will be descriptively summarized on the safety population. Previous and concomitant procedures will be summarized in the same way using MedDRA dictionary v19.0.

Therapies and procedures ongoing at the baseline visit or starting after the baseline visit will be summarized in concomitant therapies /procedures and those ending at baseline or before will be summarized in previous therapies / procedures.

#### 7.2.4 Compliance

Non-Compliance is defined as subjects who have a deviation of more than 20% from the planned 42 applications (i.e. less than 34 applications or more than 50 applications).


## 7.2.5 Statistical analysis for efficacy

A type I error of 0.05 (two-sided test) will be used to declare statistical significance.

All efficacy variables will be summarized by treatment at each visit. The categorical variables (e.g. IGA), and their changes from Baseline will be summarized by frequency and percentage for each response category (N, %). The continuous variables (EASI, objective SCORAD, TSS, and their change or percent changes, Pruritus [weekly average NRS and the VRS] and their changes from Baseline) will be summarized using means, medians, Q1, Q3, minimum, maximum, and standard deviations.

The Primary efficacy endpoint, the change from Baseline to Week 6 of the EASI score, will be analyzed using an analysis of covariance (ANCOVA) with the Treatment group as factor and Analysis center as a cofactor and EASI score at baseline as a covariate. The p-value for the treatment comparison, estimate of the Least Square means (LSmeans) treatment difference (CD5024 – Vehicle), will be generated from the ANCOVA model.

The change from Baseline in EASI score at any other evaluation visit, will be analyzed using analysis of covariance with the Treatment group as factor, Analysis center as a cofactor and EASI score at baseline as a covariate. The p- value for the treatment comparison, estimate of the LSmeans treatment difference (CD5024 – Vehicle), will be generated from the ANCOVA model.

Percent change from Baseline in EASI score at each evaluation visit will be analyzed by a CMH test stratified by analysis center with the ridit transformation and the row mean score difference statistic (FREQ procedure from SAS).

Modified objective SCORAD and TSS least square mean percent change from Baseline at each evaluation visit, will be analyzed individually using analysis of variance with the Treatment group as factor and analysis center as a cofactor.

Distribution of individual scores and their changes from Baseline, will be analyzed at each evaluation visit using the Cochran-Mantel-Haenszel (CMH) test stratified by analysis center with the ridit transformation and the row mean score difference statistic (FREQ procedure from SAS).

Proportion of subjects achieving success (IGA=0 [clear] or IGA=1 [Almost clear]) will be analyzed at each evaluation visit using the CMH test stratified by analysis center with the ridit transformation and the general association statistic (FREQ procedure from SAS).

Change in Pruritus (Weekly average NRS based on at least 4 daily scores and the VRS) will be separately analyzed at each evaluation visit by the CMH test stratified by analysis center with the ridit transformation and the row mean difference statistic (FREQ procedure from SAS).


#### 7.2.6 Statistical and analytical issues

#### 7.2.6.1 Adjustment for covariates

NA.

## 7.2.6.2 Handling of dropouts or missing data

For the primary endpoint (change from Baseline in EASI score) several sensitivity analyses will be conducted in ITT population:

- The primary imputation method will use the LOCF (Last observation carried forward) approach.
- For sensitivity purpose, the method of imputation for missing data will be MI (Multiple Imputation) using the Missing At Random (MAR) assumption. The MI procedure of the SAS system will be used to generate five sets of data with missing values imputed from observed data. It is expected that the pattern of missing data will be monotonic, with slight deviations being corrected by the Markov Chain Monte Carlo (MCMC) method of the MI procedure. Linear regression will be employed to model the missing EASI score, with the following covariates included in the imputation model: treatment and non-missing data from earlier timepoints. The imputed datasets will be analyzed using the methodology described for change from Baseline in EASI score. The results from the analysis of the multiple imputed datasets will be combined by the MIANALYZE procedure of the SAS system. The seed number to be used will be the protocol number (109696).

For secondary endpoints the LOCF method will be used.

#### 7.2.6.3 Interim analyses and data monitoring

NA

#### 7.2.6.4 Multicenter studies

Analysis center will be defined during the blind review meeting and will be included as a cofactor in the inferential analyses of primary and secondary endpoints.

## 7.2.6.5 Multiple comparison/multiplicity

The primary purpose is to compare CD5024 cream 0.3% QD daily to its vehicle in terms of EASI score. P-values for secondary criteria will be given for indicative purposes, so no adjustment will be made. All tests will be two-sided and significance will be declared at a 5% two-sided level.

Statistical Analysis Plan


#### 7.2.6.6 Use of a subset of patients

The protocol deviations will be identified during the blind review, and some of them will lead to the exclusion of the subjects from the PP analyses. PP analyses will be performed on primary and secondary endpoints.

## 7.2.6.7 Active-Control studies intended to show equivalence

NA.

## 7.2.6.8 Examination of Subgroups

Subgroup analyses will be explored by IgE on the primary endpoint. A threshold will be defined during the blind review.

## 7.3 Safety analysis

#### 7.3.1 Extent of exposure

#### 7.3.1.1 Treatment duration

Treatment duration will be calculated as the difference in days between the date of last application of medication and the date of first use + 1 during Period A. Date of last visit under treatment will be used if the date of last use is not available.

## 7.3.1.2 Quantity of product used

All collected and weighed packaging of product will be used to determine the quantity of product used per subject. Total Medication usage (g) and Daily medication usage (g/day) will be summarized by descriptive statistics. The variables will be derived by the following:

- Total medication used = total dispensed weight (g) total returned weight (g)
- Daily medication used = total medication used (g) / treatment duration (day)

As the subject will be instructed by a member of the staff on how to measure the prescribed dose using fingertip units (FTU), FTU will be summarized the same way as the medication used, Total and Daily FTU.

Statistical Analysis Plan




## 7.3.3 Laboratory parameters

For each parameter, shift tables presenting: pre-treatment (the value obtained closest and prior to the first application, in case of retest) versus Day 22 and Day 43/Early termination (last post-baseline value on treatment) will be generated. The number and percentage of subjects below, within, and above the laboratory reference ranges will be summarized. The percentage will be based on the number of subjects with data available for both pre-treatment and post-treatment.

Descriptive statistics (n, mean, min, max and median) will be performed for pre-treatment value, Day 22 and Day 43/Early termination. Change from baseline to Day 22 and to Day 43/Early termination value will also be summarized.

The maximal value will be imputed for any laboratory values below the limit of quantification (e.g. "X" will be used for "<X").

In case a parameter would a value '>X' no imputation will be made and no mean and standard deviation will be output as for IgE and Creatinine Clearance. For Creatinine Clearance the analysis will be summarized in categories:

| Creatinine Clearance |
|---------------------------------|
| > 90 mL/min/1.73m² |
| 60-89 mL/min/1.73m <sup>2</sup> |
| 30-59 mL/min/1.73m <sup>2</sup> |
| 15-29 mL/min/1.73m <sup>2</sup> |
| <15 mL/min/1.73m² |

#### 7.3.4 Vital signs, physical findings and other observations related to safety

Vital signs, physical examination and ECG will be descriptively summarized.

Statistical Analysis Plan




## 7.5 Analysis visit definition

If multiple measurements are taken in the same interval, the one closest to the target study day will be used for the analysis. If two measurements are taken with equal differences in timing compared with the target date, the nominal visit number (recorded on the CRF page) will be used. Analysis visit will apply to the summaries and analyses of all efficacy variables.

| Analysis Visit | Analysis Visit number | Target<br>Study Day | Visit Window (Study Day) |
|---|---|---|---|
| Baseline | Baseline | 1 | [≤1] |
| Week 1 | Week 1 | 8 | [2-11] |
| Week 2 | Week 2 | 15 | [12 – 18] |
| Week 3 | Week 3 | 22 | [19 – 25] |
| Week 4 | Week 4 | 29 | [26 – 32] |
| Week 5 | Week 5 | 36 | [33 – 39] |
| Week 6 | Week 6 | 43 | [40 - 46] |

Statistical Analysis Plan


#### 8 CHANGES FROM THE PROTOCOL ANALYSIS PLAN

The initial analysis plan was to perform an ANOVA on the percent change from baseline to week 6 in EASI score, but one observation appears to deviate markedly from others (200% increase of the EASI score). This outlier skews the distribution and for the intended analysis (ANOVA) increases the residual error and thus makes the statistical test less powerful and less appropriate.

Then, the change from Baseline in EASI score at Week 6 will be the primary endpoint and will be analyzed via an ANCOVA with treatment as factor, analysis center as a cofactor and EASI at Baseline as covariate. This analysis will be conducted on ITT-LOCF, ITT-MI and PP population.

Percent change from baseline at any scheduled visits will be secondary and will be analyzed via a CMH test using RIDIT transformation and row mean score statistics. This analysis will be conducted on ITT-LOCF and PP population.

#### 9 TABLES, FIGURES, AND GRAPHS

#### 9.1 Study subject

Table 9.1.1 Enrolment by country and investigator

| | CD5024 | Vehicle |
|--------------|--------|---------|
| Overall | XX | XX |
| 5xxx-PR. XXX | XX | XX |
| 5yyy-PR. YYY | XX | XX |

**Table 9.1.2** Reason for discontinuation

| | CD5024 | Vehicle |
|-------------------|------------|------------|
| N (%) | xx | XX |
| Normal Completion | xx (x.xx%) | xx (x.xx%) |
| Adverse Event | xx (x.xx%) | xx (x.xx%) |
| Subject's Request | xx (x.xx%) | xx (x.xx%) |
| Lost to Follow-up | xx (x.xx%) | xx (x.xx%) |
| Other | xx (x.xx%) | xx (x.xx%) |

Statistical Analysis Plan 

 Table 9.1.3
 Demographic data

| | | CD5024 | Vehicle |
|----------------|---------|-------------|-------------|
| N | | XX | xx |
| Gender | Female | xx(xx.x%) | xx(xx.x%) |
| | Male | xx(xx.x%) | xx(xx.x%) |
| Race | White | xx(xx.x%) | xx(xx.x%) |
| | | xx(xx.x%) | xx(xx.x%) |
| Age (in Years) | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx | XX |
| | Min;Max | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx |

 Table 9.1.4
 Baseline disease characteristics

| | | CD5024 | Vehicle |
|--------------|----------------|-------------|-------------|
| IGA | N | XX | XX |
| | 0-Clear | xx (xx.x%) | xx(xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx(xx.x%) |
| | 2-Mild | xx (xx.x%) | xx(xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx(xx.x%) |
| | 4-Severe | xx (xx.x%) | xx(xx.x%) |
| Hand IGA | N | xx | XX |
| | 0-Clear | xx (xx.x%) | xx(xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx(xx.x%) |
| | 2-Mild | xx (xx.x%) | xx(xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx(xx.x%) |
| | 4-Severe | xx (xx.x%) | xx(xx.x%) |
| BSA | N | xx | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx | XX |
| | Min;Max | XX ; XX | XX;XX |
| | Q1;Q3 | xx ; xx | xx ; xx |
| BSA affected | N | XX | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |
| | Q1;Q3 | XX ; XX | XX;XX |
| EASI | N | XX | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX | XX |
| | Min;Max | XX ; XX | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx |

Statistical Analysis Plan 

| | | CD5024 | Vehicle |
|---|---|---|---|
| Modified SCORAD | N | XX | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx |
| VRS | N | xx | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx | XX |
| | Min;Max | xx ; xx | XX ; XX |
| | Q1;Q3 | xx ; xx | XX ; XX |
| NRS | N | xx | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx | XX |
| | Min;Max | XX ; XX | XX ; XX |
| | Q1;Q3 | xx ; xx | xx ; xx |
| TSS | N | xx | XX |
| | Mean±SD | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx |
| Erythema | N | XX | XX |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx (xx.x%) |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) |
| Induration / Papulation | N | · | · |
| mudration / Fapulation | 0-Clear | XX | XX |
| | | xx (xx.x%) | xx (xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx (xx.x%) |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) |
| Oozing / Crusting | N | XX | XX |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx (xx.x%) |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) |
| Excoriation | N | XX | XX |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | ` , |
| | | · | xx (xx.x%) |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) |

Statistical Analysis Plan


| | | CD5024 | Vehicle |
|-----------------|----------------|------------|------------|
| Lichenification | N | xx | XX |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) |
| | 1-Almost Clear | xx (xx.x%) | xx (xx.x%) |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) |

# Table 9.1.5 Dataset analyzed

| | CD5024 | Vehicle | Total |
|-------------------|------------|------------|------------|
| Screened subjects | - | - | XX |
| ITT population | xx (x.xx%) | xx (x.xx%) | xx (x.xx%) |
| PP population | xx (x.xx%) | xx (x.xx%) | xx (x.xx%) |
| Safety population | xx (x.xx%) | xx (x.xx%) | xx (x.xx%) |
| PK set | xx (x.xx%) | xx (x.xx%) | xx (x.xx%) |

# **Table 9.1.6** Medical history

| | | CD5024 | Vehicle |
|-----------------|-------|------------|------------|
| Medical History | N (%) | xx | xx |
| | Yes | xx (xx.x%) | xx (xx.x%) |
| | No | xx (xx.x%) | xx (xx.x%) |

# **Table 9.1.7** Previous therapies

| | | CD5024 | | | Vehicle | |
|---|---|---|---|---|---|---|
| | n<br>therapies | n subjects | % subj. | n<br>therapies | n<br>subjects | % subj |
| Subjects with at least one previous therapy* | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| ATC Text#1 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | xx.x | XX.X | XX.X | XX.X | xx.x | XX.X |
| ATC Text#2 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | xx.x | XX.X | XX.X | XX.X | xx.x | XX.X |
| Preferred term #3 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| ATC Text#3 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | xx.x | XX.X | XX.X | XX.X | xx.x | XX.X |
| Preferred term #2 | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| ATC Text#x | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X |

<sup>\*</sup>Multiple reports by each subject are possible

Statistical Analysis Plan


**Table 9.1.8** Concomitant therapies

| | | CD5024 | | Vehicle | | |
|---|---|---|---|---|---|---|
| | n<br>therapies | n subjects | % subj. | n<br>therapies | n<br>subjects | % subj. |
| Subjects with at least one concomitant therapy* | xx.x | XX.X | xx.x | xx.x | xx.x | XX.X |
| ATC Text#1 | xx.x | XX.X | XX.X | xx.x | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | xx.x | XX.X | XX.X | xx.x | xx.x | XX.X |
| ATC Text#2 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | xx.x | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| ATC Text#3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #2 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| ATC Text#x | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

<sup>\*</sup>Multiple reports by each subject are possible

**Table 9.1.9 Summary of Previous Procedures and Non-Drug Therapies** 

| | | CD5024 | | Vehicle | | |
|---|---|---|---|---|---|---|
| | n<br>procedure<br>s | n<br>subjects | %<br>subj. | n<br>procedure<br>s | n<br>subjects | %<br>subj. |
| Subjects with at least one previous procedures and non drug therapy* | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| SOC#1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC#2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC#3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC #x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

<sup>\*</sup>Multiple reports by each subject are possible

Statistical Analysis Plan


Table 9.1.10 Summary of concomitant Procedures and Non-Drug Therapies

| | CD5024 | | | Vehicle | | |
|---|---|---|---|---|---|---|
| | n<br>procedure<br>s | n<br>subjects | %<br>subj. | n<br>procedure<br>s | n<br>subjects | %<br>subj. |
| Subjects with at least one concomitant procedures and non drug therapy* | XX.X | xx.x | XX.X | XX.X | xx.x | XX.X |
| SOC#1 | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| Preferred term #1 | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC#2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | xx.x | XX.X | XX.X | xx.x |
| Preferred term #2 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC#3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #1 | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X |
| Preferred term #2 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Preferred term #3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SOC #x | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

<sup>\*</sup>Multiple reports by each subject are possible

Table 9.1.11 Subject with major protocol deviations

| | CD5024 | | Vehicle | |
|---|---|---|---|---|
| | N<br>subj.* | %<br>subj | N<br>subj.* | %<br>subj |
| AT LEAST ONE MAJOR DEVIATION* | xx | XX.X | xx | XX.X |
| entrance criteria deviations (at baseline) | х | X.X | х | X.X |
| concomitant therapies taken during the study | х | X.X | х | X.X |
| | х | X.X | х | X.X |

<sup>\*</sup> Subjects with at least one major deviation

Numbers in columns cannot be added because a given subject may have reported more than one deviation

Table 9.1.12 Compliance

| | C | CD5024 | | icle |
|-----------------------|------------|-----------|-------------|-----------|
| | N<br>subj. | %<br>subj | N<br>subj.* | %<br>subj |
| <34 applications | x | X.X | х | X.X |
| 34 to 50 applications | x | X.X | х | X.X |
| >50 applications | x | X.X | х | X.X |

Statistical Analysis Plan


# 9.2 Efficacy analysis

## 9.2.1 Primary efficacy endpoint

 $\frac{Table \ 9.2.1.1 \ Descriptive \ results \ of \ the \ change \ from \ baseline \ in \ EASI \ score \ at \ each}{\underline{timepoint-ITT-LOCF}}$ 

| | | C | D5024 | <u>Ve</u> | <u>hicle</u> |
|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Raw Data | Change from baseline |
| <u>Baseline</u> | <u>N</u> | XX | | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | | xx.x ±xx | |
| | <u>Median</u> | <u>xx</u> | | XX | |
| | Min;Max | xx;xx | | <u>xx ; xx</u> | |
| | Q1;Q3 | xx;xx | | <u>xx ; xx</u> | |
| Day 8-LOCF | <u>N</u> | XX | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | <u>xx.x ±xx</u> | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | <u>xx</u> | <u>xx</u> | <u>xx</u> | <u>xx</u> |
| | Min;Max | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> |
| | Q1;Q3 | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> |
| Day 15-LOCF | <u>N</u> | XX | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | <u>xx.x ±xx</u> | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | <u>XX</u> | <u>xx</u> | XX |
| | Min;Max | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> |
| | Q1;Q3 | xx;xx | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> |
| Day 22-LOCF | <u>N</u> | <u>xx</u> | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | XX | XX | XX |
| | Min;Max | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> |
| | Q1;Q3 | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | XX;XX |
| Day 29-LOCF | <u>N</u> | XX | <u>XX</u> | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | <u>xx.x ±xx</u> | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | <u>XX</u> | <u>xx</u> | XX |
| | Min;Max | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | XX;XX |
| | Q1;Q3 | xx;xx | xx;xx | XX;XX | xx;xx |

Statistical Analysis Plan


| | | C | D5024 | Veh | icle |
|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Raw Data | Change from baseline |
| Day 36-LOCF | <u>N</u> | XX | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | XX | XX | XX |
| | Min;Max | xx ; xx | XX;XX | <u>xx ; xx</u> | <u>xx ; xx</u> |
| | Q1;Q3 | xx;xx | XX;XX | XX;XX | <u>xx ; xx</u> |
| Day 43-LOCF | <u>N</u> | XX | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | XX | XX | XX |
| | Min;Max | xx;xx | XX;XX | XX;XX | <u>xx ; xx</u> |
| | Q1;Q3 | xx;xx | xx;xx | xx;xx | xx;xx |

<u>Table 9.2.1.2 Statistical analysis of the change from baseline in score EASI at each timepoint – ITT-LOCF</u>

| | | CD5024 | <u>Vehicle</u> | CD5024- Vehicle |
|---|---|---|---|---|
| <u>Baseline</u> | N | xx | xx | = |
| | <u>Mean</u> | xx | xx | XX |
| | <u>SD</u> | XX | XX | XX |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 8-LOCF | N | XX | XX | = |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 15-LOCF | <u>N</u> | XX | XX | = |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 22-LOCF | <u>N</u> | XX | XX | = |
| | <u>LS-Mean</u> | <u>xx</u> | <u>xx</u> | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |

Statistical Analysis Plan


| | | CD5024 | <u>Vehicle</u> | CD5024- Vehicle |
|---|---|---|---|---|
| Day 29-LOCF | N | XX | XX | = |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | <u>xx</u> | XX |
| | p-value (1) | XX | <u>xx</u> | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | <u>xx</u> | XX |
| Day 36-LOCF | <u>N</u> | <u>xx</u> | <u>xx</u> | |
| | LS-Mean | XX | <u>xx</u> | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 43-LOCF | <u>N</u> | <u>xx</u> | XX | Ξ |
| | LS-Mean | <u>xx</u> | XX | XX |
| | <u>SE</u> | <u>xx</u> | <u>xx</u> | XX |
| | p-value (1) | <u>xx</u> | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | <u>xx</u> | XX | xx |
| | Upper bound 95%CI | XX | <u>xx</u> | <u>xx</u> |

(1) p-values from the ANCOVA model include treatment, analysis center and baseline EASI scores

<u>Table 9.2.1.3 Statistical analysis of the change from baseline in score EASI at each timepoint – ITT-MI</u>

| | | CD5024 | <u>Vehicle</u> | CD5024- Vehicle |
|---|---|---|---|---|
| <u>Baseline</u> | N | XX | XX | = |
| | <u>Mean</u> | XX | XX | XX |
| | <u>SD</u> | XX | XX | XX |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 8-MI | N | XX | XX | = |
| | <u>LS-Mean</u> | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 15-MI | <u>N</u> | XX | XX | _ |
| | <u>LS-Mean</u> | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |

Statistical Analysis Plan 

| | | CD5024 | Vehicle | CD5024- Vehicle |
|-----------|-------------------|-----------|---------|-----------------|
| Day 22-MI | N | xx | xx | = |
| | LS-Mean | XX | XX | xx |
| | <u>SE</u> | <u>xx</u> | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | xx |
| Day 29-MI | <u>N</u> | XX | XX | = |
| | <u>LS-Mean</u> | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 36-MI | N | XX | XX | = |
| | <u>LS-Mean</u> | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 43-MI | <u>N</u> | XX | XX | = |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |

(1) p-values from the ANCOVA model include treatment, analysis center and baselineEASI scores

Statistical Analysis Plan


<u>Table 9.2.1.4 Descriptive results of the change from baseline in EASI score at each timepoint – PP population</u>

| | | C | D5024 | Ve | <u>hicle</u> |
|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Raw Data | Change from baseline |
| Baseline | N | XX | | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | | xx.x ±xx | |
| | <u>Median</u> | XX | | XX | |
| | Min;Max | xx ; xx | | XX;XX | |
| | Q1;Q3 | xx ; xx | | XX;XX | |
| Day 8-PP | <u>N</u> | XX | XX | XX | XX |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | XX | XX | XX | XX |
| | Min;Max | xx ; xx | XX;XX | XX;XX | XX;XX |
| | Q1;Q3 | xx;xx | XX;XX | XX;XX | XX;XX |
| ay 15-PP | <u>N</u> | xx | XX | xx | XX |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | XX.X ±XX |
| | <u>Median</u> | xx | XX | xx | XX |
| | Min;Max | xx;xx | xx;xx | xx ; xx | XX;XX |
| | Q1;Q3 | xx ; xx | xx;xx | xx ; xx | xx;xx |
| ay 22-PP | <u>N</u> | XX | XX | XX | xx |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | xx | XX | xx | XX |
| | Min;Max | xx;xx | xx;xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;xx | xx;xx | xx ; xx | xx ; xx |
| ay 29-PP | N | xx | XX | xx | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | xx | XX | xx | xx |
| | Min;Max | xx;xx | xx;xx | xx;xx | xx;xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| ay 36-PP | N | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | XX | XX | XX |
| | Min;Max | xx ; xx | xx ; xx | XX;XX | XX ; XX |
| | Q1;Q3 | xx;xx | xx ; xx | xx ; xx | xx ; xx |
| Day 43-LOCF | N N | xx | XX | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | <u>Median</u> | <u></u> | XX | xx | XX |
| | Min;Max | xx;xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;xx | xx ; xx | xx ; xx | xx ; xx |

Statistical Analysis Plan


<u>Table 9.2.1.5 Statistical analysis of the change from baseline EASI at each timepoint – PP population</u>

| | | CD5024 | <u>Vehicle</u> | CD5024- Vehicle |
|---|---|---|---|---|
| <u>Baseline</u> | N | XX | xx | = |
| | <u>Mean</u> | XX | XX | XX |
| | <u>SD</u> | XX | XX | XX |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | xx | XX | XX |
| Day 8-PP | <u>N</u> | XX | XX | <u>=</u> |
| | LS-Mean | xx | XX | XX |
| | <u>SE</u> | xx | XX | XX |
| | p-value (1) | XX | xx | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 15-PP | <u>N</u> | XX | XX | <u>=</u> |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 22-PP | <u>N</u> | XX | XX | = |
| | LS-Mean | XX | xx | XX |
| | <u>SE</u> | XX | xx | XX |
| | p-value (1) | XX | xx | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | xx | XX |
| Day 29-PP | <u>N</u> | XX | xx | = |
| | <u>LS-Mean</u> | XX | XX | XX |
| | <u>SE</u> | XX | xx | XX |
| | p-value (1) | XX | xx | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | xx | XX |
| | Upper bound 95%CI | XX | xx | XX |

Statistical Analysis Plan


| | | CD5024 | <u>Vehicle</u> | CD5024- Vehicle |
|-----------|-------------------|--------|----------------|-----------------|
| Day 36-PP | N | XX | XX | _ |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 43-PP | N | XX | XX | _ |
| | LS-Mean | XX | XX | XX |
| | <u>SE</u> | XX | XX | XX |
| | p-value (1) | XX | XX | <u>0.xxx</u> |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |

(1) p-values from the ANCOVA model include treatment, analysis center and baseline EASI scores

<u>Table 9.2.1.6 Statistical Analysis of the percent change from baseline in EASI score at each timepoint – ITT-LOCF</u>

| | | C | D5024 | <u>Ve</u> l | nicle | <u>p-value</u> |
|---|---|---|---|---|---|---|
| | | Raw Data | Percent<br>change from<br>baseline | Raw Data | Change from baseline | |
| <u>Baseline</u> | <u>N</u> | XX | | <u>xx</u> | | |
| | <u>Mean±SD</u> | xx.x ±xx | | xx.x ±xx | | |
| | <u>Median</u> | xx | | XX | | <u>=</u> |
| | Min;Max | xx;xx | | XX;XX | | |
| | Q1;Q3 | xx ; xx | | XX;XX | | |
| Day 8-LOCF | N | xx | XX | XX | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | XX.X ±XX | xx.x ±xx | XX.X ±XX | |
| | <u>Median</u> | xx | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | xx ; xx | XX;XX | XX;XX | xx ; xx | |
| | Q1;Q3 | xx ; xx | XX;XX | XX;XX | xx ; xx | |
| Day 15-LOCF | N | xx | XX | XX | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | xx | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx;xx | XX;XX | xx;xx | |
| | Q1;Q3 | <u>xx ; xx</u> | <u>xx ; xx</u> | <u>xx ; xx</u> | xx;xx | |
| Day 22-LOCF | <u>N</u> | xx | XX | XX | XX | |
| | <u>Mean±SD</u> | XX.X ±XX | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx;xx | xx ; xx | xx;xx | xx ; xx | |

Statistical Analysis Plan


| | | CD5024 Vehicle | | <u>icle</u> | p-value | |
|---|---|---|---|---|---|---|
| | | Raw Data | Percent<br>change from<br>baseline | Raw Data | Change from baseline | |
| Day 29-LOCF | <u>N</u> | XX | <u>xx</u> | <u>xx</u> | <u>xx</u> | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | <u>xx</u> | XX | XX | <u>0.xxx</u> |
| | Min;Max | <u>xx ; xx</u> | xx;xx | xx;xx | xx;xx | |
| | Q1;Q3 | <u>xx ; xx</u> | xx;xx | xx;xx | xx;xx | |
| Day 36-LOCF | <u>N</u> | XX | XX | XX | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx ; xx | XX;XX | xx;xx | |
| | Q1;Q3 | XX;XX | xx ; xx | XX;XX | xx;xx | |
| Day 43-LOCF | <u>N</u> | XX | XX | xx | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx ; xx | xx ; xx | xx;xx | |
| | Q1;Q3 | XX;XX | xx;xx | xx ; xx | xx;xx | |

(1) p-values based on CMH test stratified by analysis center

<u>Table 9.2.1.7 Statistical Analysis results of the percent change from baseline in EASI score at each timepoint – PP</u>

| | | <u>C</u> | D5024 | <u>Ve</u> | nicle | <u>p-value</u> |
|---|---|---|---|---|---|---|
| | | Raw Data | Percent<br>change from<br>baseline | Raw Data | Change from baseline | |
| <u>Baseline</u> | <u>N</u> | XX | | XX | | |
| | <u>Mean±SD</u> | XX.X ±XX | | xx.x ±xx | | |
| | <u>Median</u> | XX | | XX | | Ξ. |
| | Min;Max | XX;XX | | XX;XX | | |
| | Q1;Q3 | XX;XX | | XX;XX | | |
| Day 8-PP | <u>N</u> | XX | XX | XX | XX | |
| | <u>Mean±SD</u> | XX.X ±XX | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | <u>xx</u> | XX | <u>xx</u> | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx;xx | XX;XX | xx;xx | |
| | Q1;Q3 | XX;XX | xx;xx | XX;XX | xx;xx | |
| <u>Day 15-PP</u> | <u>N</u> | XX | <u>xx</u> | XX | XX | |
| | <u>Mean±SD</u> | XX.X ±XX | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | xx ; xx | XX;XX | xx ; xx | |
| | Q1;Q3 | XX;XX | xx ; xx | XX;XX | xx ; xx | |

Statistical Analysis Plan 

| | | C | D5024 | <u>Ve</u> | nicle | p-value |
|---|---|---|---|---|---|---|
| | | Raw Data | Percent<br>change from<br>baseline | Raw Data | Change from baseline | |
| Day 22-PP | N | <u>xx</u> | XX | <u>xx</u> | XX | |
| | <u>Mean±SD</u> | XX.X ±XX | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | <u>xx</u> | XX | XX | <u>0.xxx</u> |
| | Min;Max | <u>xx ; xx</u> | xx;xx | XX;XX | xx;xx | |
| | Q1;Q3 | XX;XX | xx ; xx | XX;XX | xx;xx | |
| <u>Day 29-PP</u> | N | XX | <u>xx</u> | XX | XX | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | <u>xx</u> | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | <u>xx ; xx</u> | <u>xx ; xx</u> | xx;xx | |
| | Q1;Q3 | XX;XX | <u>xx ; xx</u> | <u>xx ; xx</u> | xx;xx | |
| Day 36-PP | <u>N</u> | XX | <u>xx</u> | <u>xx</u> | <u>xx</u> | |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | XX | <u>xx</u> | <u>xx</u> | <u>xx</u> | <u>0.xxx</u> |
| | Min;Max | XX;XX | XX;XX | <u>xx ; xx</u> | XX;XX | |
| | Q1;Q3 | XX;XX | xx;xx | <u>xx ; xx</u> | xx;xx | |
| Day 43-PP | <u>N</u> | <u>xx</u> | <u>xx</u> | <u>xx</u> | XX | · |
| | <u>Mean±SD</u> | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | <u>Median</u> | <u>xx</u> | XX | XX | XX | <u>0.xxx</u> |
| | Min;Max | XX;XX | <u>xx ; xx</u> | <u>xx ; xx</u> | xx;xx | |
| | Q1;Q3 | XX;XX | <u>xx ; xx</u> | <u>xx ; xx</u> | xx;xx | |

(1) p-values based on CMH test stratified by analysis center

Statistical Analysis Plan


# 9.2.2 Secondary efficacy endpoints

Table 9.2.2.1 Distribution of Investigator Global Assessment by visit –ITT LOCF

| | | CD5024 | Vehicle | p-value |
|-------------|----------------|------------|------------|---------|
| Baseline | N (%) | XX | XX | - |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| Day 8-LOCF | N (%) | XX | XX | 0.xxx |
| - | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 15-LOCF | N (%) | XX | XX | 0.xxx |
| • | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 22-LOCF | N (%) | XX | XX | 0.xxx |
| • | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 29-LOCF | N (%) | XX | XX | 0.xxx |
| • | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 36-LOCF | N (%) | XX | XX | 0.xxx |
| - | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 43-LOCF | N (%) | xx | XX | 0.xxx |
| - | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center

Statistical Analysis Plan


 $Table\ 9.2.2.2\ Distribution\ of\ Investigator\ Global\ Assessment\ by\ visit-PP$ 

| | | CD5024 | Vehicle | p-value |
|----------|----------------|------------|------------|---------|
| Baseline | N (%) | XX | XX | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| Day 8 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 15 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 22 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 29 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 36 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 43 | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center

Statistical Analysis Plan


**Table 9.2.2.3 Summary of IGA Success - ITT LOCF** 

| | | CD5024 | Vehicle | p-value |
|----------|------------|------------|------------|---------|
| Baseline | N (%) | XX | xx | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| Day 8 | N (%) | XX | xx | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |
| Day 15 | N (%) | XX | XX | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |
| Day 22 | N (%) | XX | XX | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |
| Day 29 | N (%) | XX | XX | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |
| Day 36 | N (%) | XX | XX | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |
| Day 43 | N (%) | XX | xx | 0.xxx |
| | Success | xx (xx.x%) | xx (xx.x%) | |
| | Failure | xx (xx.x%) | xx (xx.x%) | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center

## **Table 9.2.2.4 Summary of IGA Success - PP**

Table 9.2.2.5 Distribution of the Hand Investigator Global Assessment by visit –ITT LOCF

Same as for IGA

Table 9.2.2.6 Distribution of the Hand Investigator Global Assessment by visit -PP

Same as for IGA

Statistical Analysis Plan 

 $Table \ 9.2.2.7 \ Descriptive \ results \ of \ the \ TSS \ at \ each \ timepoint-ITT-LOCF$ 

| | | CD5024 | | Vehicle | | | |
|---|---|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Percent change from baseline | Raw Data | Change from baseline | Percent change from baseline |
| Baseline | N | xx | | | XX | | |
| | Mean±SD | xx.x ±xx | | | xx.x ±xx | | |
| | Median | XX | | | xx | | |
| | Min;Max | xx ; xx | | | xx ; xx | | |
| | Q1;Q3 | xx ; xx | | | xx ; xx | | |
| Day 8-LOCF | N | xx | xx | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | xx | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 15-LOCF | N | XX | xx | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | xx | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 22-LOCF | N | XX | xx | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 29-LOCF | N | XX | xx | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | xx | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 36-LOCF | N | XX | xx | xx | xx | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | XX ; XX | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | XX ; XX | xx ; xx | xx ; xx |
| Day 43-LOCF | N | XX | xx | xx | XX | xx | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | XX | xx | XX | xx | XX |
| | Min;Max | xx ; xx | XX ; XX | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;xx | xx ; xx | xx;xx | xx ; xx | xx;xx | xx ; xx |

Statistical Analysis Plan


Table 9.2.2.8 Statistical analysis of the percent change from baseline of the TSS at each timepoint – ITT-LOCF

| | | CD5024 | Vehicle | CD5024- Vehicle |
|-------------|-------------------|--------|---------|-----------------|
| Baseline | N | xx | xx | - |
| | Mean | xx | XX | XX |
| | SD | xx | XX | XX |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | xx | XX |
| Day 8-LOCF | N | XX | xx | - |
| | LS-Mean | XX | xx | XX |
| | SE | XX | xx | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | xx | XX |
| | Upper bound 95%CI | XX | xx | XX |
| Day 15-LOCF | N | XX | XX | - |
| • | LS-Mean | XX | XX | XX |
| | SE | XX | xx | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 22-LOCF | N | XX | XX | - |
| • | LS-Mean | XX | XX | xx |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 29-LOCF | N | XX | xx | - |
| • | LS-Mean | XX | XX | XX |
| | SE | XX | XX | XX |
| | p-value (1) | XX | xx | 0.xxx |
| | Lower bound 95%CI | XX | xx | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 36-LOCF | N | XX | xx | - |
| • | LS-Mean | XX | XX | xx |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%Cl | XX | XX | XX |
Statistical Analysis Plan


| | | CD5024 | Vehicle | CD5024- Vehicle |
|-------------|-------------------|--------|---------|-----------------|
| Day 43-LOCF | N | XX | XX | - |
| | LS-Mean | XX | XX | XX |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | xx | xx |

<sup>(1)</sup> p-values from the ANOVA model including treatment and analysis center effects

Table 9.2.2.9 Descriptive results of the TSS at each timepoint – PP population

Table 9.2.2.10 Statistical analysis of the percent change from baseline of the TSS at each timepoint – PP

Table 9.2.2.11 Descriptive results of the Modified Objective SCORAD at each timepoint – ITT population

| | | | CD5024 | | | Vehicle | |
|---|---|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Percent change from baseline | Raw Data | Change from baseline | Percent<br>change from<br>baseline |
| Baseline | N | XX | | | xx | | |
| | Mean±SD | xx.x ±xx | | | xx.x ±xx | | |
| | Median | XX | | | XX | | |
| | Min;Max | xx ; xx | | | xx ; xx | | |
| | Q1;Q3 | xx ; xx | | | xx ; xx | | |
| Day 8-LOCF | N | XX | xx | xx | XX | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | XX | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 15-LOCF | N | XX | xx | xx | XX | xx | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | XX | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 22-LOCF | N | XX | xx | xx | XX | XX | xx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | xx | xx |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | XX;XX | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |

Statistical Analysis Plan


| | | | CD5024 | | | Vehicle | |
|---|---|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Percent change from baseline | Raw Data | Change from baseline | Percent change from baseline |
| Day 29-LOCF | N | XX | XX | xx | XX | xx | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | xx | XX |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 36-LOCF | N | XX | XX | xx | XX | xx | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | XX | xx | XX | xx | XX |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| Day 43-LOCF | N | XX | XX | xx | XX | xx | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx |
| | Median | XX | xx | xx | XX | XX | XX |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |

Table 9.2.2.12 Statistical analysis of the percent change from baseline of the Modified Objective SCORAD at each timepoint – ITT-LOCF

| | | CD5024 | Vehicle | CD5024- Vehicle |
|-------------|-------------------|--------|---------|-----------------|
| Baseline | N | xx | xx | - |
| | Mean | xx | xx | xx |
| | SD | xx | xx | xx |
| | Lower bound 95%CI | xx | xx | xx |
| | Upper bound 95%CI | xx | xx | xx |
| Day 8-LOCF | N | xx | xx | - |
| | LS-Mean | xx | xx | xx |
| | SE | xx | XX | xx |
| | p-value (1) | xx | xx | 0.xxx |
| | Lower bound 95%CI | xx | XX | xx |
| | Upper bound 95%CI | xx | xx | xx |
| Day 15-LOCF | N | xx | xx | - |
| | LS-Mean | xx | xx | xx |
| | SE | xx | xx | xx |
| | p-value (1) | xx | xx | 0.xxx |
| | Lower bound 95%CI | xx | XX | XX |
| | Upper bound 95%CI | XX | xx | XX |

Statistical Analysis Plan


| | | CD5024 | Vehicle | CD5024- Vehicle |
|-------------|-------------------|--------|---------|-----------------|
| Day 22-LOCF | N | XX | xx | - |
| | LS-Mean | XX | xx | XX |
| | SE | XX | xx | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | xx | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 29-LOCF | N | XX | XX | - |
| | LS-Mean | XX | xx | XX |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 36-LOCF | N | XX | XX | - |
| | LS-Mean | XX | XX | XX |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |
| Day 43-LOCF | N | XX | XX | - |
| | LS-Mean | XX | XX | XX |
| | SE | XX | XX | XX |
| | p-value (1) | XX | XX | 0.xxx |
| | Lower bound 95%CI | XX | XX | XX |
| | Upper bound 95%CI | XX | XX | XX |

<sup>(1)</sup> p-values from the ANOVA model including treatment and analysis center effects

Table 9.2.2.13 Descriptive results of the Modified Objective SCORAD at each timepoint – PP population

Table 9.2.2.14 Statistical analysis of the percent change from baseline of the Modified Objective SCORAD at each timepoint – PP

Statistical Analysis Plan


 $Table\ 9.2.2.15\ Distribution\ of\ Erythema\ score\ by\ visit\ -ITT\ LOCF$ 

| | | CD5024 | Vehicle | p-value |
|-------------|----------------|------------|------------|---------|
| Baseline | N (%) | XX | XX | • |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 8-LOCF | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 15-LOCF | N (%) | XX | XX | 0.xxx |
| | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 22-LOCF | N (%) | XX | XX | 0.xxx |
| - | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 29-LOCF | N (%) | XX | XX | 0.xxx |
| - | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 36-LOCF | N (%) | XX | XX | 0.xxx |
| • | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |
| Day 43-LOCF | N (%) | XX | XX | 0.xxx |
| ÷ | 0-Clear | xx (xx.x%) | xx (xx.x%) | |
| | 1-Almost clear | xx (xx.x%) | xx (xx.x%) | |
| | 2-Mild | xx (xx.x%) | xx (xx.x%) | |
| | 3-Moderate | xx (xx.x%) | xx (xx.x%) | |
| | 4-Severe | xx (xx.x%) | xx (xx.x%) | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center, for the change from baseline

Statistical Analysis Plan


Table 9.2.2.16 Distribution of Erythema score by visit – PP

Table 9.2.2.17 Distribution of Induration/Papulation score by visit – ITT LOCF

Table 9.2.2.18 Distribution of Induration/Papulation score by visit – PP

Table 9.2.2.19 Distribution of Oozing/Crusting score by visit – ITT LOCF

Table 9.2.2.20 Distribution of Oozing/Crusting score by visit – PP

**Table 9.2.2.21 Distribution of Excoriation score by visit – ITT LOCF** 

Table 9.2.2.22 Distribution of Excoriation score by visit – PP

Table 9.2.2.23 Distribution of Lichenification score by visit – ITT LOCF

Table 9.2.2.24 Distribution of Lichenification score by visit – PP

Statistical Analysis Plan


Table 9.2.2.25 Descriptive results of the weekly average NRS at each timepoint – ITT population

| | | C | D5024 | Ve | hicle | p-value(1) |
|---|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Raw Data | Change from baseline | |
| Baseline | N | xx | | xx | | |
| | Mean±SD | xx.x ±xx | | xx.x ±xx | | |
| | Median | xx | | xx | | |
| | Min;Max | xx ; xx | | xx ; xx | | |
| | Q1;Q3 | xx ; xx | | xx ; xx | | |
| Week 1 - LOCF | N | xx | XX | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | xx | XX | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| Week 2-LOCF | N | xx | xx | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | xx | xx | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| Week 3 -LOCF | N | xx | xx | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | xx | XX | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| Week 4 -LOCF | N | xx | XX | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | xx | xx | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| Week 5 -LOCF | N | xx | xx | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | XX | xx | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| Week 6 -LOCF | N | XX | xx | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | XX | xx | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center Baseline is the mean of the values collected from Day -1 to Day -3

Statistical Analysis Plan


## Table 9.2.2.26 Descriptive results of the weekly average NRS at each timepoint – PP population

Table 9.2.2.27 Descriptive results of the VRS at each timepoint – ITT population

| | | C | D5024 | Vel | hicle | p-value(1) |
|---|---|---|---|---|---|---|
| | | Raw Data | Change from baseline | Raw Data | Change from baseline | |
| Baseline | N | xx | | xx | | |
| | Mean±SD | xx.x ±xx | | xx.x ±xx | | |
| | Median | XX | | xx | | |
| | Min;Max | xx ; xx | | xx ; xx | | |
| | Q1;Q3 | xx ; xx | | xx ; xx | | |
| Day 43 -LOCF | N | xx | xx | xx | xx | 0.xxx |
| | Mean±SD | xx.x ±xx | xx.x ±xx | xx.x ±xx | xx.x ±xx | |
| | Median | xx | xx | xx | xx | |
| | Min;Max | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |
| | Q1;Q3 | xx ; xx | xx ; xx | xx ; xx | xx ; xx | |

<sup>(1)</sup> p-values based on CMH test stratified by analysis center

Table 9.2.2.28 Descriptive results of the VRS at each timepoint – PP population

Statistical Analysis Plan


# 9.2.3 Subgroup analyses

Table 9.2.3.1 Descriptive results of EASI at each timepoint broken down by IgE- ITT population

| | | | | lgE | <x< th=""><th></th><th></th><th colspan="4">IgE&gt;=X</th></x<> | | | IgE>=X | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | CD502 | 4 | | Vehicle | Э | | CD502 | 4 | | Vehicle | ) |
| | | Raw<br>Data | Change<br>from<br>baselin<br>e | Percent<br>change<br>from<br>baselin<br>e | Raw<br>Data | Change<br>from<br>baselin<br>e | Percent<br>change<br>from<br>baselin<br>e | Raw<br>Data | Change<br>from<br>baselin<br>e | Percent<br>change<br>from<br>baselin<br>e | Raw<br>Data | Change<br>from<br>baselin<br>e | Percent<br>change<br>from<br>baselin<br>e |
| Baselin | N | XX | | xx | | | | | | | XX | | |
| е | Mean±SD | xx.x<br>±xx | | xx.x<br>±xx | | | | | | | xx.x<br>±xx | | |
| | Median | XX | | XX | | | | | | | XX | | |
| | Min;Max | xx;<br>xx | | xx ; xx | | | | | | | xx;<br>xx | | |
| | Q1;Q3 | xx;<br>xx | | xx ; xx | | | | | | | xx;<br>xx | | |
| Day 8- | N | XX | XX | xx | XX | xx | xx | XX | XX | xx | XX | XX | XX |
| LOCF | Mean±SD | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | xx | xx | xx | xx | xx | XX | XX | xx | XX | xx | xx |
| | Min;Max | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx;xx | xx ; xx |
| | Q1;Q3 | xx;<br>xx | xx ; xx | xx;xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx;xx | xx ; xx |
| Day 15- | N | XX | xx | xx | XX | XX | xx | XX | XX | xx | XX | XX | XX |
| LOCF | Mean±SD | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | XX | xx | XX | xx | xx | XX | XX | xx | XX | XX | XX |
| | Min;Max | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx;xx | xx ; xx |
| | Q1;Q3 | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx;xx | xx ; xx |
| Day 22- | N | XX | XX | xx | XX | XX | XX | XX | XX | xx | XX | XX | XX |
| LOCF | Mean±SD | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | XX.X<br>±XX | XX.X<br>±XX | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | xx | xx | XX | XX | XX | XX | XX | xx | XX | XX | XX |
| | Min;Max | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | XX;<br>XX | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |

Statistical Analysis Plan 

| | | | | lgE | <x< th=""><th></th><th></th><th></th><th></th><th>lgE</th><th>&gt;=X</th><th></th><th></th></x<> | | | | | lgE | >=X | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | CD502 | 4 | | Vehicle | Э | | CD502 | 4 | | Vehicle | ) |
| Day 29- | N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| LOCF | Mean±SD | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Min;Max | XX;<br>XX | xx ; xx | xx ; xx | XX;<br>XX | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx; | xx ; xx | xx ; xx | xx; | xx ; xx | xx ; xx | xx; | xx ; xx | xx ; xx | xx; | xx ; xx | xx ; xx |
| | | XX | | | XX | | | XX | | | XX | | |
| Day 36-<br>LOCF | N | XX | XX | XX | XX | XX | XX | XX | XX | xx | XX | XX | xx |
| | Mean±SD | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Min;Max | XX;<br>XX | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |
| Day 43- | N | XX | XX | xx | XX | xx | XX | XX | XX | XX | XX | XX | xx |
| LOCF | Mean±SD | XX.X<br>±XX | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx | XX.X<br>±XX | xx.x<br>±xx | xx.x<br>±xx | xx.x<br>±xx |
| | Median | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | Min;Max | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx;xx | xx;xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |
| | Q1;Q3 | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx | xx;<br>xx | xx ; xx | xx ; xx |

Statistical Analysis Plan


# 9.3 Safety analysis

### 9.3.1 Extent of exposure

Table 9.3.1.1 Treatment applications- Safety population

| | | CD5024 | Vehicle |
|------------------------------|---------|----------|----------|
| Treatment duration (in days) | N | xx | XX |
| ( · · · <b>,</b> · , | Mean±SD | xx.x ±xx | xx.x ±xx |
| | Median | xx | XX |
| | Min;Max | xx ; xx | xx ; xx |

# Table 9.3.1.2 Quantity of product used (g)

| | | CD5024 | Vehicle |
|-------------------------------|---------|----------|----------|
| Total medication used (g) | N | XX | XX |
| | Mean±SD | xx.x ±xx | XX.X ±XX |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |
| Daily medication used (g/day) | N | XX | XX |
| | Mean±SD | xx.x ±xx | XX.X ±XX |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |

# Table 9.3.1.3 Quantity of product applied in Fingertips unit (FTU)

| | | CD5024 | Vehicle |
|----------------------------------|---------|----------|----------|
| Total number of fingertips (FTU) | N | XX | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |
| Daily fingertips (FTU/day) | N | XX | XX |
| | Mean±SD | xx.x ±xx | xx.x ±xx |
| | Median | XX | XX |
| | Min;Max | xx ; xx | xx ; xx |

Protocol No: RD.03.SPR.109696 Statistical Analysis Plan 

| CCI |
|-----|

Protocol No: RD.03.SPR.109696 Statistical Analysis Plan 



Protocol No: RD.03.SPR.109696 Statistical Analysis Plan 



Statistical Analysis Plan




# 9.3.3 Laboratory parameters

# 9.3.3.1 Blood chemistry

Table 9.3.3.1.1 Blood chemistry shift table

| | | | | | | Baseline | е | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | CD50 | )24 | | | Veh | icle | |
| | | | Low | Normal | High | Missing | Low | Normal | High | Missing |
| Day 22 | Parameter#1 | Low | - | x (x.x) | - | - | - | - | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | ٠ | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | ٠ | - |
| | | Missing | - | - | - | - | - | x (x.x) | ٠ | - |
| | Parameter#2 | Low | - | x (x.x) | - | - | - | x (x.x) | ٠ | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | • | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | - | - | - | - | | - | - |
| Day 43/early<br>Termination | Parameter#1 | Low | - | - | - | - | - | - | • | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | Parameter#2 | Low | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | • | - |
| | | Missing | - | - | - | - | - | - | • | - |
| | | | | | - | - | - | | - | - |

Statistical Analysis Plan 

Table 9.3.3.1.2 Blood chemistry parameter over time

| | | | CD | 5024 | Veh | icle |
|---|---|---|---|---|---|---|
| | | | Raw data | Change | Raw data | Change |
| Parameter# | Baseline | N | xx | | XX | |
| 1 | | Mean±SD | x.xx±x.xx | | x.xx±x.xx | |
| | | Median | x.xx | | X.XX | |
| | | Min;Max | x.xx;x.xx | | x.xx;x.xx | |
| Day 22 | Day 22 | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |
| Da | Day 43 / Early Termination | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |
| Parameter# | Baseline | N | xx | | XX | |
| 2 | | Mean±SD | x.xx±x.xx | | x.xx±x.xx | |
| | | Median | x.xx | | X.XX | |
| | | Min;Max | x.xx;x.xx | | x.xx;x.xx | |
| | Day 22 | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | x.xx |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |
| | Day 43 / Early Termination | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | x.xx |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |

Statistical Analysis Plan 

### 9.3.3.2 Hematology

Table 9.3.3.2.1 Hematology shift table

| | | | | | | Baseline | • | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | CD50 | )24 | | | Veh | icle | |
| | | | Low | Normal | High | Missing | Low | Normal | High | Missing |
| Day 22 | Parameter#1 (unit) | Low | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | - | - | - | - | | - | - |
| | Parameter#2 (unit) | Low | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | - | - | - | - | - | - | - |
| Day 43/Early<br>Termination | Parameter#1 (unit) | Low | - | -x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | | - | - | - | | - | - |
| | Parameter#2 (unit) | Low | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | - | - | - | - | - | - | - |
| | | | | | - | - | - | | - | - |

Statistical Analysis Plan


**Table 9.3.3.2.2 Descriptive analysis for Creatinine Clearance** 

| | | CD5024 | Vehicle |
|---|---|---|---|
| Baseline | > 90 mL/min/1.73m² | x (x.x) | x (x.x) |
| | 60-89 mL/min/1.73m <sup>2</sup> | x (x.x) | x (x.x) |
| | 30-59 mL/min/1.73m <sup>2</sup> | x (x.x) | x (x.x) |
| | 15-29 mL/min/1.73m² | x (x.x) | x (x.x) |
| | <15 mL/min/1.73m² | x (x.x) | x (x.x) |
| Day 22 | > 90 mL/min/1.73m² | x (x.x) | x (x.x) |
| | 60-89 mL/min/1.73m² | x (x.x) | x (x.x) |
| | 30-59 mL/min/1.73m² | x (x.x) | x (x.x) |
| | 15-29 mL/min/1.73m² | x (x.x) | x (x.x) |
| | <15 mL/min/1.73m² | x (x.x) | x (x.x) |
| Day 43/Early Termination | > 90 mL/min/1.73m² | x (x.x) | x (x.x) |
| | 60-89 mL/min/1.73m² | x (x.x) | x (x.x) |

Table 9.3.3.2.3 Hematology parameter over time

| | | | CD | 5024 | Veh | icle |
|---|---|---|---|---|---|---|
| | | | Raw data | Change | Raw data | Change |
| Parameter#1 | Baseline | N | xx | | XX | |
| | | Mean±SD | x.xx±x.xx | | x.xx±x.xx | |
| | | Median | x.xx | | X.XX | |
| | | Min;Max | x.xx;x.xx | | x.xx;x.xx | |
| | Day 22 | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | X.XX;X.XX | -x.xx;x.xx |
| | Day 43 / Early Termination | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |

Statistical Analysis Plan 

| | | | CD | 5024 | Veh | icle |
|---|---|---|---|---|---|---|
| | | | Raw data | Change | Raw data | Change |
| Parameter#2 | Baseline | N | xx | | XX | |
| | | Mean±SD | x.xx±x.xx | | x.xx±x.xx | |
| Day | | Median | x.xx | | X.XX | |
| | | Min;Max | x.xx;x.xx | | x.xx;x.xx | |
| | Day 22 | N | xx | XX | XX | xx |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |
| | Day 43 / Early Termination | N | xx | XX | XX | xx |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |

### 9.3.3.3 Coagulation

Table 9.3.3.3.1 Coagulation shift table

| | | | | Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | CD5024 | | | Vehicle | | | |
| | | | Low | Normal | High | Missing | Low | Normal | High | Missing |
| Day 22 | Prothrombin<br>Ratio | Low | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | - | - | - | - | | | - |
| Day 43/Early<br>Termination | Prothrombin<br>Ratio | Low | - | x (x.x)- | - | - | - | x (x.x) | - | - |
| | | Normal | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | High | - | x (x.x) | - | - | - | x (x.x) | - | - |
| | | Missing | - | | - | _ | - | | - | - |

Statistical Analysis Plan


Table 9.3.3.3.2 Coagulation parameter over time

| | | | CD | 5024 | Veh | icle |
|---|---|---|---|---|---|---|
| | | | Raw data | Change | Raw data | Change |
| Prothrombin | Baseline | N | xx | | XX | |
| Ratio Day 22 | Mean±SD | x.xx±x.xx | | x.xx±x.xx | | |
| | | Median | x.xx | | X.XX | |
| | | Min;Max | x.xx;x.xx | | x.xx;x.xx | |
| | Day 22 | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |
| | Day 43 / Early Termination | N | xx | XX | XX | XX |
| | | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | | Median | x.xx | X.XX | X.XX | X.XX |
| | | Min;Max | x.xx;x.xx | -x.xx;x.xx | x.xx;x.xx | -x.xx;x.xx |

## 9.3.4 Vital Sign and physical examination and other information related to safety

Table 9.3.4.1 Descriptive results of vital signs

| | | | CD5024 | | | Vehicle | |
|---|---|---|---|---|---|---|---|
| | | Systolic<br>blood<br>pressure<br>(mmHg) | Diastolic<br>blood<br>pressure<br>(mmHg) | Pulse rate<br>(bpm) | Systolic<br>blood<br>pressure<br>(mmHg) | Diastolic<br>blood<br>pressure<br>(mmHg) | Pulse rate<br>(bpm) |
| Baseline | N | xx | XX | xx | XX | XX | xx |
| | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | Median | X.XX | X.XX | x.xx | X.XX | X.XX | x.xx |
| | Min;Max | x.xx;x.xx | x.xx;x.xx | x.xx;x.xx | x.xx;x.xx | x.xx;x.xx | x.xx;x.xx |
| | N | xx | xx | xx | xx | xx | xx |
| | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | Median | x.xx | X.XX | x.xx | X.XX | X.XX | x.xx |
| | Min;Max | x.xx;x.xx | x.xx;x.xx | x.xx;x.xx | X.XX;X.XX | x.xx;x.xx | x.xx;x.xx |
| Day 54/Early | N | xx | XX | xx | XX | XX | xx |
| termination | Mean±SD | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx | x.xx±x.xx |
| | Median | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Min;Max | x.xx;x.xx | x.xx;x.xx | X.XX;X.XX | X.XX;X.XX | x.xx;x.xx | x.xx;x.xx |

Statistical Analysis Plan


Table 9.3.4.2 Descriptive results of physical examination

| | | CD5024 | Vehicle |
|---|---|---|---|
| Baseline | N (%) | XX | xx |
| | Normal Physical Examination | xx (xx.x) | xx (xx.x) |
| Day 15 | N (%) | xx | XX |
| | Normal Physical Examination | xx (xx.x) | xx (xx.x) |
| | Ex #1 Neurological Function | x (x.x) | x (x.x) |
| | Ex #2 Skin | x (x.x) | x (x.x) |
| Day 29 | N (%) | XX | XX |
| | Normal Physical Examination | xx (xx.x) | xx (xx.x) |
| | Ex #1 Neurological Function | x (x.x) | x (x.x) |
| | Ex #2 Skin | | |
| | | x (x.x) | x (x.x) |
| Day 43 | N (%) | XX | XX |
| | Normal Physical Examination | xx (xx.x) | xx (xx.x) |
| | Ex #1 Neurological Function | x (x.x) | x (x.x) |
| | Ex #2 Skin | x (x.x) | x (x.x) |
| Day 54/Early termination | N (%) | XX | XX |
| | Normal Physical Examination | xx (xx.x) | xx (xx.x) |
| | Ex #1 Neurological Function | x (x.x) | x (x.x) |
| | Ex #2 Skin | x (x.x) | x (x.x) |

Table 9.3.4.3 Descriptive results of ECG

| | | CD5024 | Vehicle |
|--------------------------|----------|-----------|-----------|
| Baseline | N (%) | xx | XX |
| | Normal | xx (xx.x) | xx (xx.x) |
| | Abnormal | xx (xx.x) | xx (xx.x) |
| Day 43/Early termination | N (%) | xx | XX |
| | Normal | xx (xx.x) | xx (xx.x) |
| | Abnormal | x (x.x) | x (x.x) |

Protocol No: RD.03.SPR.109696 Statistical Analysis Plan 

